CLINICAL TRIAL: NCT02442518
Title: Antenatal Diagnosis of Placental Attachment Disorders
Acronym: ADoPAD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: NICOLA FRATELLI (Other)
Collaborators: Azienda Ospedaliera San Gerardo di Monza (Other); IRCCS Burlo Garofolo (Other); Azienda Ospedaliera Ospedali Riuniti Villa Sofia Cervello (Other); Azienda Ospedaliero-Universitaria di Parma (Other); ARNAS Civico di Cristina Benefratelli, Palermo (Unknown); Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other); University of Milan (Other); A.O.U. Città della Salute e della Scienza (Other); Ospedale Valduce, Como (Unknown); Azienda Ospedaliera Bolognini di Seriate Bergamo (Other)
Responsible Party: Sponsor-Investigator, NICOLA FRATELLI, MD, Università degli Studi di Brescia
Organization: Università degli Studi di Brescia (Other)
Other Study IDs: 1837
Record Dates: First submitted 2015-04-20; First posted 2015-05-13 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Placenta Accreta; Placenta Previa
Keywords: placenta accreta; placenta previa; ultrasound
MeSH Terms: conditions — Placenta Accreta; Placenta Previa

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — histopathological samples from women with placenta previa diagnosed with ultrasound in the 3rd trimester of pregnancy
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- women with placenta praevia: women with placenta previa diagnosed at antenatal ultrasound in the third trimester of pregnancy (lower placental edge within 20 mm from the internal os above 26 week's gestation)
  Interventions: Procedure: antenatal ultrasound

INTERVENTIONS:
Procedure: antenatal ultrasound — Transabdominal and Transvaginal ultrasound examinations were performed in the third trimester (with some fluid in the bladder so that the uterine bladder interface could be evaluated well).

SUMMARY:
The accuracy of sonographic prenatal detection of invasive placentation is unclear. The objective of this prospective, multicenter, observational study is to assess the performance of ultrasound for prenatal identification of invasive placentation in women with placenta previa.

This study involves more than 25 hospitals in Italy.

DETAILED DESCRIPTION:
Background: Morbidly adherent placenta is a spectrum of conditions characterized by an abnormal adherence of the placenta to the implantation site. Three major variants of adherent placentation can be recognized according to the degree of trophoblastic invasion through the myometrium and the uterine serosa: placenta accreta, placenta increta and placenta percreta. All varieties of invasive placentation are associated with a significant increase in maternal morbidity.Placenta previa and previous uterine surgery represent the major risk factors for invasive placentation. Prenatal diagnosis of invasive placentation is associated with a reduced risk of maternal complications such as peripartum blood loss, need for transfusions and rate of hysterectomy, as it allows a preplanned treatment of the condition, however the performance of antenatal ultrasound and of different sonographic signs is not consistent across published studies because of limited sample size, retrospective design, variability of inclusion criteria and definition of invasive placentation.

Objectives: The aim of this study is to systematically assess the performance of ultrasound in the prenatal diagnosis of placenta accreta and its variants and to evaluate the role of the different specific ultrasound signs in predicting disorders of invasive placentation. The sonographic signs assessed in this study were: (1) vascular lacunae within the placenta, (2) loss of normal hypoechoic retroplacental zone, (3) interruption of the bladder line and/or focal exophytic masses extending into the bladder space, considered together and labeled as 'abnormalities of the uterus - bladder interface.

Design:prospective, multicenter, observational study of pregnant women with placenta previa.

Methods: The investigators hypothesized that ultrasound has a sensitivity of at least 80% and a specificity of at least 97%, with 10% confidence intervals, for antenatal diagnosis of invasive placentation.The investigators would require 2048 women with placenta previa, of whom approximately 61 (3%) will have morbidly adherent placenta, to test the null hypothesis with a 0.05 risk of type I error (alpha). Supposing a 10% of women with incomplete follow up the investigators aim to enroll 2254 women in this study.

Diagnostic criteria that suggested placenta accreta, increta, or percreta included one or more of the following situations: (1) obliteration of the clear space, defined as the obliteration of any part of the echolucent area located between the uterus and placenta; (2) visualization of placental lacunae, defined as multiple linear, irregular vascular spaces within the placenta; and (3) interruption of the posterior bladder wall-uterine interface such that the usual continuous echolucent line appears instead as a series of dashes.

The degree of placental invasion was defined as follows: (i) placenta accreta was assumed when placental 'cones' disrupted the decidual zone with mildly increased vascularization around these cones ; (ii) placenta increta was diagnosed when placental invasion into the myometrium was sonographically suspected as a result of the presence of irregular and diffuse demarcation of the placental - uterine wall interface and thinning of the myometrium that was overlying the placental - myometrial tissue. Placenta increta was also characterized by increased vascularization and irregularly shaped intraplacental vascular lacunae, resembling the characteristic 'moth damage' appearance ; and (iii) the sonographic finding of placenta percreta was defined by a complete absence of the myometrium, with the placenta extending to the serosa, or beyond, including vascular breakthrough.In addition, placenta percreta was also characterized by massive subplacental hypervascularization, with vessels extending irregularly into the placental - myometrial tissue and with numerous large intraplacental lacunae.

Clinical and histopathological assessment of placental invasion:

Sonographic findings were compared with the clinical outcome during and after delivery and the histomorphological examination of the placenta, performed by pathologists experienced in obstetric histopathology, who were blinded to the sonographic findings.

..........................................................................................................

Main Outcomes measure:

Primary Outcome: sensitivity (SN), specificity(SP), positive likelihood ratio (LR+), negative likelihood ratio (LR - ) and diagnostic odds ratio (DOR) of antenatal ultrasound and different sonographic signs for in prediction of morbidly adherent placenta.

Secondary Outcome: to evaluate whether the maximum degree of placental invasion (placenta accreta, increta or percreta) can be predicted with antenatal ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Placenta previa diagnosed with ultrasound above 26 weeks' gestation (lower edge reached and/or overlapped the internal cervical os, or the lower edge was between 0.1 and 20.0 mm from the internal cervical os)

Exclusion Criteria:

* Age < 18 years
* prepartum bleeding or fetal distress requiring immediate emergency Cesarean section before the enrollment of the woman

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women with placenta previa diagnosed at antenatal ultrasound in the third trimester of pregnancy (lower placental edge within 20 mm from the internal os above 26 week's gestation)
Sampling Method: Non-Probability Sample
Enrollment: 2254 (Estimated)
Dates: Start 2015-02; Primary Completion 2018-03 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
diagnostic accuracy of sonographic prenatal detection of invasive placentation | clinical and histopathological assessment of placental invasion at delivery

SECONDARY OUTCOMES:
maximum degree of placental invasion | clinical and histopathological assessment of placental invasion at delivery

CONTACTS AND LOCATIONS:
Overall Officials: NICOLA FRATELLI, MD, Principal Investigator — BRESCIA UNIVERSITY, SPEDALI CIVILI DI BRESCIA; GIUSEPPE CALI, MD, Principal Investigator — ARNAS Civico di Cristina Benefratelli
Locations (3):
- Italy (3):
  - Brescia University, Spedali Civili Di Brescia, Brescia, Brescia
  - Azienda Ospedaliera San Gerardo di Monza, Monza, MB
  - ARNAS CIVICO di Cristina Benefratelli, Palermo, Palermo

REFERENCES:
- [Background] Fitzpatrick KE, Sellers S, Spark P, Kurinczuk JJ, Brocklehurst P, Knight M. The management and outcomes of placenta accreta, increta, and percreta in the UK: a population-based descriptive study. BJOG. 2014 Jan;121(1):62-70; discussion 70-1. doi: 10.1111/1471-0528.12405. Epub 2013 Aug 7. PMID 23924326
- [Background] Fitzpatrick KE, Sellers S, Spark P, Kurinczuk JJ, Brocklehurst P, Knight M. Incidence and risk factors for placenta accreta/increta/percreta in the UK: a national case-control study. PLoS One. 2012;7(12):e52893. doi: 10.1371/journal.pone.0052893. Epub 2012 Dec 27. PMID 23300807
- [Background] Warshak CR, Ramos GA, Eskander R, Benirschke K, Saenz CC, Kelly TF, Moore TR, Resnik R. Effect of predelivery diagnosis in 99 consecutive cases of placenta accreta. Obstet Gynecol. 2010 Jan;115(1):65-69. doi: 10.1097/AOG.0b013e3181c4f12a. PMID 20027036
- [Background] Tan CH, Tay KH, Sheah K, Kwek K, Wong K, Tan HK, Tan BS. Perioperative endovascular internal iliac artery occlusion balloon placement in management of placenta accreta. AJR Am J Roentgenol. 2007 Nov;189(5):1158-63. doi: 10.2214/AJR.07.2417. PMID 17954654
- [Background] Eller AG, Porter TF, Soisson P, Silver RM. Optimal management strategies for placenta accreta. BJOG. 2009 Apr;116(5):648-54. doi: 10.1111/j.1471-0528.2008.02037.x. Epub 2009 Feb 4. PMID 19191778
- [Background] Dilauro MD, Dason S, Athreya S. Prophylactic balloon occlusion of internal iliac arteries in women with placenta accreta: literature review and analysis. Clin Radiol. 2012 Jun;67(6):515-20. doi: 10.1016/j.crad.2011.10.031. Epub 2012 Jan 2. PMID 22218410
- [Background] D'Antonio F, Iacovella C, Bhide A. Prenatal identification of invasive placentation using ultrasound: systematic review and meta-analysis. Ultrasound Obstet Gynecol. 2013 Nov;42(5):509-17. doi: 10.1002/uog.13194. Epub 2013 Oct 2. PMID 23943408
- [Background] Chalubinski KM, Pils S, Klein K, Seemann R, Speiser P, Langer M, Ott J. Prenatal sonography can predict degree of placental invasion. Ultrasound Obstet Gynecol. 2013 Nov;42(5):518-24. doi: 10.1002/uog.12451. Epub 2013 Oct 9. PMID 23471888
- [Background] Oppenheimer L; MATERNAL FETAL MEDICINE COMMITTEE. RETIRED: Diagnosis and management of placenta previa. J Obstet Gynaecol Can. 2007 Mar;29(3):261-266. doi: 10.1016/S1701-2163(16)32401-X. PMID 17346497
- [Background] Comstock CH. Antenatal diagnosis of placenta accreta: a review. Ultrasound Obstet Gynecol. 2005 Jul;26(1):89-96. doi: 10.1002/uog.1926. PMID 15971281
- [Background] Cali G, Giambanco L, Puccio G, Forlani F. Morbidly adherent placenta: evaluation of ultrasound diagnostic criteria and differentiation of placenta accreta from percreta. Ultrasound Obstet Gynecol. 2013 Apr;41(4):406-12. doi: 10.1002/uog.12385. PMID 23288834
- [Background] Bossuyt PM, Reitsma JB, Bruns DE, Gatsonis CA, Glasziou PP, Irwig LM, Lijmer JG, Moher D, Rennie D, de Vet HC; Standards for Reporting of Diagnostic Accuracy. Towards complete and accurate reporting of studies of diagnostic accuracy: the STARD initiative. Standards for Reporting of Diagnostic Accuracy. Clin Chem. 2003 Jan;49(1):1-6. doi: 10.1373/49.1.1. PMID 12507953
- [Background] Wortman AC, Alexander JM. Placenta accreta, increta, and percreta. Obstet Gynecol Clin North Am. 2013 Mar;40(1):137-54. doi: 10.1016/j.ogc.2012.12.002. PMID 23466142
- [Background] Jones SR, Carley S, Harrison M. An introduction to power and sample size estimation. Emerg Med J. 2003 Sep;20(5):453-8. doi: 10.1136/emj.20.5.453. PMID 12954688